CLINICAL TRIAL: NCT03474315
Title: Interactive Patient's Assistant to Optimize Long-term Care in Patients With Chronic Health Failure and Determine Which Parameters of CIED Indicate the Requirement for Ambulatory Follow-up
Brief Title: Interactive Patient's Assistant - LUCY
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Marcin Grabowski, Clinical Professor, Medical University of Warsaw
Other Study IDs: LUCY
Record Dates: First submitted 2017-12-13; First posted 2018-03-22 (Actual); Last update posted 2018-03-22 (Actual); Status verified 2018-03

CONDITIONS: Chronic Heart Failure
Keywords: Cardiac implantable electronic device; Cardiac resynchronization therapy; Implantable cardioverter-defibrillator; Machine learning; Mobile application; Patient's assistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- CHF and CIED patients: 600 CHF patients with ICD or CRT admitted to regulatory ambulatory visit.
  Interventions: Diagnostic Test: Multivariate assessment

INTERVENTIONS:
Diagnostic Test: Multivariate assessment — Patient's status assessment according to clinical evaluation and data acquired from the implanted device.

SUMMARY:
Patients with chronic heart failure (CHF) and reduced left ventricle ejection fraction benefit from cardiac resynchronization therapy (CRT) and implantable cardioverter defibrillator (ICD). Currently used devices, besides delivering low and high-energy therapies, record patient's activity and many hemodynamic parameters. However, increasing numbers of patient with CRT and ICD devices produce overload of cardiology centers where patients are admitted to ambulatory visits. Contrarily, there are technological possibilities for remote monitoring proven to be effective in recognizing damage of the implanted device and risk of exacerbation of chronic heart failure. Patients' registries show that majority of ambulatory visits are unproductive and do not result in significant modification of device's parameters. Promising experiences with application of data mining and machine learning techniques allow us to assume probable benefits from using modern methods of data analysis in determination of requirement for ambulatory follow-up on basis of data gathered through telemonitoring and clinical assessment of a patient.

Aim of the study is to find multivariate model predicting the requirement for ambulatory follow-up of IECD.

ELIGIBILITY:
Inclusion Criteria:

* 18-90 years old
* Chronic heart failure (NYHA class I to III)
* Implanted ICD or CRT (at least 30 days before inclusion)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be consisted of one patient group: 600 CHF patients with implanted ICD or CRT admitted to regulatory ambulatory visit.
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2018-04 (Estimated); Primary Completion 2019-02 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Ambulatory visit qualified as meaningful due to change in pharmacotherapy or ICD parameters related to tachycardia detection or treatment. | 1 day
  Primary outcome is composed of:
  * any change in pharmacotherapy (modification of agents or doses) related to patient's clinical status assessed during the visit,
  * any change in tachyarrythmia counter or discriminator status,
  * any change in tachyarrythmia threshold,
  * ventricular undersensing or oversensing.

SECONDARY OUTCOMES:
Ambulatory visit qualified as meaningful due to alarming condition related to ICD. | 1 day
  Secondary outcome is composed of:
  * sustained or treated ventricular tachyarrythmia,
  * any not previously diagnosed supraventricular tachyarrythmia,
  * elective replacement indicator,
  * atrial undersensing or oversensing,
  * atrial or ventricular ineffective pacing.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Medical Informatics and Telemedicine, Warsaw, Masovian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No